CLINICAL TRIAL: NCT01562470
Title: Clinical Trial to Assess the Efficacy and Safety of a Novel Cellulite Cream in Reducing the Appearance of Cellulite in Human Subjects
Brief Title: Clinical Trial to Assess the Efficacy and Safety of a Novel Cellulite Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-104-002
Record Dates: First submitted 2011-08-16; First posted 2012-03-23 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Thigh Cellulite
Keywords: cellulite; reduction; cream; thighs; women
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- herbal-based cellulite cream (Experimental): Trial subjects will apply the treatment cream to one thigh and placebo to the other thigh, by random allocation.
  Interventions: Other: Cellulite reduction cream

INTERVENTIONS:
Other: Cellulite reduction cream — 1/8 tsp cellulite cream will be applied to the thigh twice daily - in the morning and at night, for a period of 16 weeks.

SUMMARY:
Study Hypothesis: That the test product will reduce thigh cellulite more that the placebo.

This will be a double-blind, placebo-controlled study involving subjects with distinctive cellulite appearance on both thighs. Subjects will apply test cream to one thigh and placebo to the other, by random allocation, and cellulite appearance will be measured at week 0, 8 and 16. Cellulite photographs will also be assessed by a (study blinded) trial researcher, who will assess cellulite appearance on a precisely-measured upper leg area. The subjects' own perception of cellulite appearance, from their diaries, will be numerically coded, and all three measures will be collated and analysed statistically.

DETAILED DESCRIPTION:
Twenty subjects will be recruited through advertisements in local newspapers. Eligible subjects will be asked to visit the lab, where they will sign an information/consent form and answer a series of questions to determine their eligibility. If eligible, each subject will be asked to have their upper leg cellulite photographed, and thigh circumference will be measured. They will be given two containers of cream, labelled R (for right thigh) and L (for left thigh) which have been pre-weighed in their containers, and they will be instructed on how to apply the cream. They will record their perception of the amount of cellulite on a weekly basis, and they will also record any adverse events. At the two and four-month time-points, they will return to the lab with their diaries and cream. The cream in its container will be weighed to ensure compliance, and the diaries will be examined and returned to the participants. Thighs will again be photographed and circumference measured. At the four-month visit, subjects will return any remaining product for weighing, as well as their diaries for analysis.

Photographs from each subject will be coded and cellulite marks assessed by arranging the photographs chronologically, i.e. timepoint 1, timepoint 2 and timepoint 3. They will also be assessed by a (blinded) trial researcher, who will assess cellulite appearance on a precisely-measured upper leg area in the photographs. The subjects' own perception of cellulite appearance, from their diaries, will be numerically coded, and all three measures will be collated and analysed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 years
* Cellulite present equally on both thighs
* Willing to apply cream, as directed, for 16 weeks
* Willing to maintain habitual diet throughout the trial
* Willing to refrain from making any lifestyle changes during the life of the trial (exercise regimes, specific diets or cleanses)
* Will to refrain from making any changes to smoking habits during the study period
* Participant is in good health on the basis of medical history
* Participant understands the study procedures and provides informed consent (signed) to participate and authorizes the release of relevant protected health information to the study investigators

Exclusion Criteria:

* Use of medications known to influence cellulite appearance
* Any leg surgical visit scheduled during trial
* Known intolerance or sensitivity to any ingredients in the study product
* Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
thigh cellulite appearance | 16 weeks
  Reduction of cellulite appearance, as assessed by photographs, self-assessment and clinician assessment.

SECONDARY OUTCOMES:
Uper leg circumference and fat content | 16 weeks
  Reduction of upper leg circumference as measured by cm tape measure, and reduction of fat content of upper leg as measured using fat calipers
Presence/absence of adverse reactions | 16 weeks
  Any incidence of an adverse event or events will be recorded in an Adverse Events Diary, and results collated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Traplin, MD, Study Director — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.; Maggie Laidlaw, Ph.D., Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource Diagnostics Inc., Guelph, Ontario, Canada